CLINICAL TRIAL: NCT01249573
Title: The Effect of Fascia Therapy and Transcutaneous Fibrolysis on Acute Ankle Sprain in Young Adults.
Brief Title: The Effect of Fascia Therapy and Transcutaneous Fibrolysis on Acute Ankle Sprain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Prof. Dr. Philip Roosen, University Ghent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC/2010/580
Record Dates: First submitted 2010-10-20; First posted 2010-11-30 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Acute Ankle Distortion
Keywords: fascia therapy; transcutaneous fibrolysis; acute ankle distortion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- fascia therapy (Experimental): arm where fascia therapy is used as a treatment for an acute ankle distortion
  Interventions: Other: fascia therapy or transcutaneous fibrolysis
- transcutaneous fibrolysis (Experimental): arm where transcutaneous fibrolysis is used as a treatment for an acute ankle distortion
  Interventions: Other: fascia therapy or transcutaneous fibrolysis
- placebo (Placebo Comparator): arm where placebo therapy is used as a treatment for an acute ankle distortion
  Interventions: Other: fascia therapy or transcutaneous fibrolysis

INTERVENTIONS:
Other: fascia therapy or transcutaneous fibrolysis — fascia therapy or transcutaneous fibrolysis as treatment for an acute ankle distortion

SUMMARY:
This study investigates the immediate effect of fascia therapy and transcutaneous fibrolysis in the treatment of an acute ankle sprain. These treatments will be compared to a placebo group.

DETAILED DESCRIPTION:
Ankle sprain is the most occurring sport related injury. In spite of the high prevalence of this injury and the often residual symptoms, there is a large variety in diagnostic approach and therapeutic protocols. Concerning the treatment of an acute ankle sprain, it remains a challenge to minimize injury consequences on short and long term.

In this study we investigate the immediate effect of two therapeutic techniques: fascia therapy and transcutaneous fibrolysis. They will be compared to a third group, who receives a placebo treatment. Muscle strength, muscle vascularisation, muscle tenderness and joint position sense are measured before and after treatment.

The purpose of this study is to contribute to the knowledge of treating acute ankle sprains.

ELIGIBILITY:
Inclusion Criteria:

* acute ankle sprain

Exclusion Criteria:

* none

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
effect of fascia therapy | baseline measurements and within 1 hour after treatment
  The effect of fascia therapy on an acute ankle distortion. Measurement of muscle power, muscle saturation, joint position sense, tenderness and disability questionnaires.

SECONDARY OUTCOMES:
complaints registration | baseline, 1 hour after treatment and 3 days later
  Self-assessed complaints registration.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Roosen, Prof, PhD, Principal Investigator — University Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium